CLINICAL TRIAL: NCT03654534
Title: Oral Nutritional Supplements Compared With Standard Diet in Postoperative Gastric Cancer Patients With Adjuvant Chemotherapy: a Multicenter, Open-label, Phase 3 Randomised Controlled Trial
Brief Title: Oral Nutritional Supplements Compared With Standard Diet in Postoperative Gastric Cancer Patients With Adjuvant Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Zhiwei, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCCGPS3
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; chemothrapy; oral nutritional supplements; malnutrition
MeSH Terms: conditions — Stomach Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oral nutritional supplements (Experimental): NutrenOpimum administration was recommended with a dosage of 400 kcal/400 ml per day within 7 days postoperatively and was continued for 3 months postoperatively.
  Interventions: Dietary Supplement: NutrenOpimum
- standard diet (No Intervention): The control group was given no additional postoperative nutritional supplementation (standard diet).

INTERVENTIONS:
Dietary Supplement: NutrenOpimum — NutrenOpimum administration was recommended with a dosage of 400 kcal/400 ml per day within 7 days postoperatively and was continued for 3 months postoperatively.
  Arms: oral nutritional supplements

SUMMARY:
Background: It is known that postoperative malnutrition remains inevitable for gastric cancer patients with adjuvant chemotherapy, which could have prejudicial influence on the compliance of subsequent adjuvant chemotherapy and survival of the patients. A multi-institutional prospective phase 2 study had demonstrated the efficacy of oral nutritional supplements (ONS) for gastric cancer patients undergoing gastrectomy. However, previous studies did not focus the gastric cancer patients with adjuvant chemotherapy. Thus, it is unknown whether the ONS could benefit the gastric cancer patients with adjuvant chemotherapy. A multicenter, phase 3 randomised controlled trial was conducted to compare the ONS with standard diet for postoperative gastric cancer patients with adjuvant chemotherapy. Patients and method: In this study, pathological confirmed stage II-III or T1N1M0 gastric cancer patients who are supposed to receive adjuvant chemotherapy, aged from 18 to 75 years, with body mass index (BMI) from 18.5 to 28.0 kg/m2, and with Eastern Cooperative Oncology Group performance status ≤2, are randomized 1:1 to receive oral administration of NutrenOpimum (Nestle Suisse S.A.), a liquid enteral nutritional food for special medical purpose (FSMP), or standard diet. NutrenOpimum administration was recommended with a dosage of 400 kcal/400 ml per day within 7 days postoperatively and was continued for 3 months postoperatively. The primary end point was postoperative malnutrition, as defined as ratio of the weight loss at 3 months postoperatively to the days 7 postoperatively body weight (body weight loss ratio) higher than 10%; body weight loss ratio at 1, 3, 6 months. Secondary end points were chemotherapy withdrawal, time to adjuvant chemotherapy failure, period of adjuvant chemotherapy, quality of life, grade 3/4 neutropenia, thrombocytopenia, anemia, and severe side effects on digestive tract. Final study analysis will be conducted after the last patient's enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. be proven to be primary adenocarcinoma of gastric cancer and pathological confirmed stage II-III or T1N1M0
2. age: 18-75 years
3. Eastern Cooperative Oncology Group performance status: 0~2
4. body mass index: 18.5-28.0kg/m2
5. able to ingest semiliquid diet
6. without other malignancies with exception of the cured cervical carcinoma in situ and basal cell carcinoma
7. anticipated overall survival time ≥ 6 months
8. anticipated period of adjuvant chemotherapy ≥ 3
9. without severe mental disorder
10. without severe digestive disease
11. without Acquired Immune Deficiency Syndrome or diabetes mellitus
12. without communication barrier
13. informed consensus of patients

Exclusion Criteria:

1. with unstable hemodynamics
2. with severe nausea or vomit which cannot be controlled by drugs
3. allergic reaction to NutrenOpimum
4. dysfunction of other organs
5. with severe disease, such as infection, stroke, heart failure or stock
6. other situation to be judged not adaptive to the study by investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-09-16 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
postoperative malnutrition | 3 months postoperatively
  the weight loss at 3 months postoperatively to the days 7 postoperatively body weight (body weight loss ratio) higher than 10%
body weight loss ratio at 1, 3, 6 months | 1,3,6 months postoperatively
  the ratio of the weight loss at 1,3,6 months postoperatively to the days 7 postoperatively body weight

SECONDARY OUTCOMES:
chemotherapy withdrawal | 6 months
  chemotherapy withdrawal by the adverse events or recurrence
time to adjuvant chemotherapy failure | 6 months
  Time to adjuvant treatment chemotherapy failure (TTF) were calculated using the Kaplan-Meier method and compared by the log-rank test
period of adjuvant chemotherapy | 6 months
  period of adjuvant chemotherapy
quality of life | 6 months
  quality of life at 1,3 and 6 months as evaluated by EORTC QLQ-C30
grade 3/4 neutropenia, thrombocytopenia, anemia | 6 months
  grade 3/4 neutropenia, thrombocytopenia, anemia during adjuvant chemotherapy
severe side effects on digestive tract | 6 months
  severe side effects on digestive tract during adjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Zhiwei Zhou, Ph.D., Study Chair — SunYat-sen University
Locations (1):
- SunYat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No